CLINICAL TRIAL: NCT02588118
Title: Effect of Gender on the Pharmacokinetics-pharmacodynamics of Propofol and Cisatracurium Besylate
Brief Title: Gender and PK-PD of Propofol and Cisatracurium
Acronym: BIS5
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Ashraf Dahaba, MD, Principle Investigator, Medical University of Graz
Other Study IDs: MUGraz5
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Gender
MeSH Terms: conditions — Coitus | interventions — Propofol; cisatracurium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- male group: Propofol 2 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 1 min (t2). Patients will be monitored using bispectral index monitoring for propofol and Relaxometer mechanomyograph neuromuscular monitoring for cisatracurium. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph for Pharmacokinetic analysis.
  Interventions: Drug: propofol; Drug: Cisatracurium
- female group: Propofol 2 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 1 min (t2). Patients will be monitored using bispectral index monitoring for propofol and Relaxometer mechanomyograph neuromuscular monitoring for cisatracurium. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph for Pharmacokinetic analysis.
  Interventions: Drug: propofol; Drug: Cisatracurium

INTERVENTIONS:
Drug: propofol — Propofol 2 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 1 min (t2). Patients will be monitored using bispectral index monitoring for propofol and Relaxometer mechanomyograph neuromuscular monitoring for cisatracurium. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph for Pharmacokinetic analysis.
  Other Names: diprivan
Drug: Cisatracurium — Propofol 2 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 1 min (t2). Patients will be monitored using bispectral index monitoring for propofol and Relaxometer mechanomyograph neuromuscular monitoring for cisatracurium. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph for Pharmacokinetic analysis.
  Other Names: nimbix

SUMMARY:
In recent years it has become clear that gender differences exist both in the pharmacokinetics and the pharmacodynamics of drugs related to the practice of anesthesia. Differences in pharmacokinetics are more straightforward to study than differences in clinical effects. However, isolated pharmacokinetic data are of less value if they are not accompanied by measurements of clinical effects. Males are more sensitive than females to propofol. It may therefore be necessary to decrease the propofol dose by 30-40% in males. Females have 20-30% greater sensitivity to the muscle relaxant effects.

DETAILED DESCRIPTION:
Background: In recent years it has become clear that gender differences exist both in the pharmacokinetics and the pharmacodynamics of drugs related to the practice of anesthesia. Differences in pharmacokinetics are more straightforward to study than differences in clinical effects. However, isolated pharmacokinetic data are of less value if they are not accompanied by measurements of clinical effects. Males are more sensitive than females to propofol. It may therefore be necessary to decrease the propofol dose by 30-40% in males. Females have 20-30% greater sensitivity to the muscle relaxant effects.

Methods: Anaesthesia is induced with propofol 2 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 1 min from propofol administration (t2). Patients will be monitored using the conventionally available bispectral index monitoring for propofol concentrations and Relaxometer mechanomyograph neuromuscular monitoring for cisatracurium. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph. Pharmacokinetic analysis was performed by fitting the cisatracurium blood concentration time profile of individual patients, to non-compartmental as well as multi-compartmental pharmacokinetic models.

ELIGIBILITY:
Inclusion Criteria:

1. either males or females

Exclusion Criteria:

1. Liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: differences between equal numbers of males and females
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
propofol elimination half life | before administration till 120 minutes
  Propofol 3 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 2 min (t2). Patients will be monitored using bispectral index monitoring for propofol. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph for Pharmacokinetic analysis.

SECONDARY OUTCOMES:
cisatracurium elimination half life | before administration till 120 minutes
  Propofol 3 mg/kg (t0) followed by cisatracurium 0.1 mg/kg 2 min (t2). Patients will be monitored using TOF-Watch neuromuscular monitoring for cisatracurium. Serial arterial blood samples (5 ml) were withdrawn in EDTA-tubes before cisatracurium administration, 1, 3, 5, 7, 10, 13, 16, 19, 22, 25, 30, 60 and 90 min following administration. Blood samples were assayed in duplicate using high performance liquid chromatograph for Pharmacokinetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Dahaba, Principal Investigator — Medical University of Graz
Locations (2):
- Medical University of Graz, Graz, Austria
- Xijing hospital of Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Schmith VD, Fiedler-Kelly J, Phillips L, Grasela TH Jr. Prospective use of population pharmacokinetics/pharmacodynamics in the development of cisatracurium. Pharm Res. 1997 Jan;14(1):91-7. doi: 10.1023/a:1012015719694. PMID 9034227
- [Background] Vuyk J, Oostwouder CJ, Vletter AA, Burm AG, Bovill JG. Gender differences in the pharmacokinetics of propofol in elderly patients during and after continuous infusion. Br J Anaesth. 2001 Feb;86(2):183-8. doi: 10.1093/bja/86.2.183. PMID 11573657